CLINICAL TRIAL: NCT03835858
Title: Safety of Airway Clearance Combined With Bronchodilator and Hypertonic Saline in Non-hospitalized Infants With Acute Viral Bronchiolitis
Brief Title: Safety of Airway Clearance in Non-hospitalized Infants With Acute Viral Bronchiolitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guadarrama Hospital (Other)
Collaborators: Fisiobronquial Clínicas (Other)
Responsible Party: Principal Investigator, J. Nicolas Cuenca Zaldivar, Rehabilitation Service Principal Investigator, Guadarrama Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6.0
Record Dates: First submitted 2019-02-07; First posted 2019-02-11 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Bronchiolitis
Keywords: Physical Therapy; Respiratory; Pediatric
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Intervention Model Description: Prospective, quasi-experimental study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Respiratory physiotherapy (Other): The protocol consists of 20 minutes of FR based on nasal washes in sitting, prolonged slow expiration: passive technique of expiratory help applied to the baby through a slow thoracic-abdominal pressure that begins at the end of a spontaneous expiration and continuing to the residual volume. The physiotherapist through the the provoked cough or stimulation of the trachea achieves the expectoration of the sputum.
  Interventions: Other: Respiratory physiotherapy

INTERVENTIONS:
Other: Respiratory physiotherapy — The protocol consists of 20 minutes of FR based on nasal washes in sitting, prolonged slow expiration: passive technique of expiratory help applied to the baby through a slow thoracic-abdominal pressure that begins at the end of a spontaneous expiration and continuing to the residual volume. The physiotherapist through the the provoked cough or stimulation of the trachea achieves the expectoration of the sputum.

SUMMARY:
Bronchiolitis is a disease that can occur in a mild form and moderate, and often does not require hospitalization. The technique of prolonged slow expiration followed by cough caused in children not hospitalized with mild and moderate bronchiolitis can improve clinical severity

DETAILED DESCRIPTION:
Once each patient legal guardians has signed the informed consent document and it has been verified that the inclusion criteria are met, it will be assigned the same identification number (ID) that is related to its Clinical History (CH) by simple coding; custody of the file with the relationship of each ID with its CH will be the responsibility of the principal investigator.

Before starting the treatment protocol, a blind evaluator treats the was assigned the patient classifies the child according to the initial score of clinical severity proposed by Wang, in addition to the measurement of SO2 and heart rate measured through a pulse oximeter.

The protocol consists of 20 minutes of FR based on nasal washes in sitting, prolonged slow expiration: passive technique of expiratory help applied to the baby through a slow thoracic-abdominal pressure that begins at the end of a spontaneous expiration and continuing to the residual volume. The physiotherapist through the provoked cough or stimulation of the trachea achieves the expectoration of the sputum.

Care must be taken during the maneuvers of maintaining a position of the infant in supine decubitus in 30 degrees of slope, to avoid episodes of gastroesophageal reflux and decrease the risk of vomiting.

They are considered as criteria of cessation of the physiotherapeutic intervention, alterations abrupt of the respiratory rhythm (brady or tachypnea), stare, ocular revulsion, hiccups or hypertonia and changes in skin color (pallor or cyanosis). In addition to these clinical manifestations, it establishes that if the father or legal guardian demands it, the application of the protocol would be terminated.

In order to evaluate the immediate effect of the protocol, which is established as the effect evaluated 10 minutes immediately after the intervention was applied, the doctor again performs a measurement of SO2, heart rate and respiratory rate, and classify again according to the criteria of Wang's clinical severity scale and anotate any adverse event. At 20 minutes the same medical evaluator performs the same assessment.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following inclusion criteria:

* Have an age between 2 months and 12 months.
* Have medical diagnosis of first episode of BQ of maximum 48 hours of evolution.
* Not previously received respiratory physiotherapy since its diagnosis.
* Have the informed consent signed by the child's legal guardians.

Exclusion Criteria:

The exclusion criteria are:

* Acute BQ with score> 9 according to the Wang clinical scale.
* Pathology associated cardiac, neurological or traumatic.
* Previous hospitalizations for wheezing.
* Medical diagnosis of recurrent sibilant.

Ages: 2 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 265 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-05-05 (Actual); Study Completion 2019-05-05 (Actual)

PRIMARY OUTCOMES:
Wang clinical severity scale | 12 weeks
  The clinical severity scale of Wang evaluates the respiratory rate, the presence of wheezing and intercostal retraction, and the patient's general condition, puncturing each dimension from 0 (the possible state) to 3 (values within normal), in addition to offer different cut points for children with more or less than 6 months.

SECONDARY OUTCOMES:
Oxygen saturation | 12 weeks
  Measured by a pulse oximeter (Radical 7 Touchscreen by Massimo®, Masimo Corporation, Irvine, CA).

CONTACTS AND LOCATIONS:
Overall Officials: J. Nicolas Cuenca Zaldivar, Principal Investigator — Guadarrama Hospital
Locations (1):
- J.Nicolas Cuenca Zaldivar, Guadarrama, Madrid, Spain